CLINICAL TRIAL: NCT06535867
Title: The Efficacy of Conventional Screening Versus mHealth Screening in Early Detection of Oral Potentially Malignant Disorders and Oral Cancer Amongst the Rural Population of Varanasi: A Prospective and Blinded Study
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 24-148
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Smoking; Smoking, Cigarette; Smoking, Tobacco; Betel Chewer's Mucosa; Tobacco Use; Tobacco Smoking; Alcohol Drinking; Smokeless Tobacco Hyperkeratosis
Keywords: smoking; smoking, cigarette; smoking, tobacco; smokeless tobacco; betel leaf; areca nut; paan masala; alcohol use; Memorial Sloan Kettering Cancer Center; 24-148
MeSH Terms: conditions — Smoking; Cigarette Smoking; Tobacco Smoking; Tobacco Use; Alcohol Drinking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants from Varanasi: Participants will be recruited from Varanasi.
  Interventions: Diagnostic Test: mHealth

INTERVENTIONS:
Diagnostic Test: mHealth — The mobile health (mHealth) program will be used for early detection of oral cancer and pre-cancer lesions, and to improve awareness of oral cancer among the population and knowledge of oral cancer diagnosis among frontline health providers.
  Other Names: Mobile Health

SUMMARY:
Mobile health (mHealth) will be used for early detection of oral cancer and pre-cancer lesions, and to improve awareness of oral cancer among the population and knowledge of oral cancer diagnosis among frontline health providers. This program is inclusive of long term surveillance to downstage oral cancer in India

ELIGIBILITY:
Inclusion Criteria:

Positive for any one or more of the following:

* All individuals aged above 18 years positive for habits (smoking and smokeless tobacco, chewing betel leaf, areca nut, paan masala, and/or regular use of alcohol)
* Clinical signs/symptoms (non-healing ulcers, white/ red/red & white patches in the mouth, restriction of mouth opening and swelling of the neck)
* All individuals aged above 40 irrespective of habit/oral lesions

Exclusion Criteria:

* Individuals already diagnosed with oral cancer and undergoing treatment for oral cancer
* Under treatment for tuberculosis or suffering from any acute illness/ debilitating systemic disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Field health personnel (FHP) with help of ASHA (a healthcare network in rural areas) will visit household and collect mobile phone numbers in Varanasi.
Sampling Method: Non-Probability Sample
Enrollment: 5122 (Estimated)
Dates: Start 2024-07-30 (Actual); Primary Completion 2031-07-30 (Estimated); Study Completion 2031-07-30 (Estimated)

PRIMARY OUTCOMES:
Comparison of mHealth with conventional oral cancer screening | Up to 5 years
  To compare the efficacy of conventional screening with mHealth in identification of oral potentially malignant disorders (OPMDs) / oral cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Milind Rajadhyaksha, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center (All protocol activites), New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org